CLINICAL TRIAL: NCT00106886
Title: HOPE-2 Study (Heart Outcomes Prevention Evaluation-2 Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Population Health Research Institute (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HOPE-2, CIHR FRN # MT-15428
Record Dates: First submitted 2005-03-31; First posted 2005-04-01 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Disease; Myocardial Infarction; Stroke; Cancer
Keywords: homocysteine; folic acid; micronutrients; multivitamins; vitamin supplements
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Neoplasms | interventions — Folic Acid; Vitamin B 6; Vitamin B 12

INTERVENTIONS:
Drug: Folic acid, vitamin B6 and B12 or placebo

SUMMARY:
The purpose of the HOPE-2 study is to determine whether long term supplementation with folic acid, vitamins B6 and B12 aimed at homocyst(e)ine reduction reduces the rates of major fatal and nonfatal cardiovascular events in patients with established cardiovascular disease and/or diabetes mellitus.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains a major cause of mortality and morbidity in most developed countries and accounts for approximately 40% of all deaths in Canada. Reductions in cholesterol, lowering of blood pressure and smoking cessation have been shown to be effective strategies in cardiovascular prevention; however, these major "classical cardiovascular risk factors" along with nonmodifiable risk factors, cannot fully explain why certain individuals develop atherosclerotic cardiovascular diseases, while others do not. Other "emerging" cardiovascular risk factors are currently under investigation. There is a large body of consistent, biologically plausible evidence linking hyperhomocyst(e)inemia to cardiovascular risk and the association is graded. A simple, nontoxic therapeutic intervention in the form of multivitamins - folic acid and vitamins B6 and B12 - has been shown to be highly effective in reducing homocyst(e)ine levels, irrespective of the underlying cause. To date, however, there are no good clinical trials evaluating the efficacy of homocyst(e)ine-lowering therapies in reducing major cardiovascular events. The impact of this simple intervention on cardiovascular morbidity and mortality remains to be demonstrated.

Study Hypothesis: Evaluate if long-term therapy with folic acid and vitamins B6 and B12 compared to placebo reduces the risk of major fatal and nonfatal cardiovascular events.

Importance of the Study: The "homocyst(e)ine theory of atherosclerosis" remains an important unanswered question in cardiovascular medicine. If indeed a combination of multivitamins is found to be effective in reducing cardiovascular events, it is expected that this safe, inexpensive and easily administered therapy would be widely used world-wide. Therefore, the results of this trial could have a significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 55 years of age or over with established CVD and at high risk for future fatal and nonfatal CV events, defined as:

  1. Documented coronary artery disease (CAD);
  2. Documented peripheral vascular disease (PVD);
  3. Documented cerebrovascular disease;
  4. Diabetes with one of the following; additional cardiovascular risk factors:

  i) hypertension (BP >160 mmHg systolic or >90 mmHg diastolic or on treatment); ii) total cholesterol >5.2 mmol/L (>200 mg/dl); iii) HDL cholesterol <0.9 mmol/L (3.5 mg/dl); iv) current cigarette smoker; v) any evidence of previous vascular disease
* Provision of informed consent

Exclusion Criteria:

* Current use of any vitamin supplements containing folic acid >200 micrograms/day. The patients taking such vitamin supplements can be asked if they agree to discontinue these supplements. If they agree, they can be randomized to the study following a one month wash-out period.
* Known previous adverse reactions to folic acid and/or vitamin B6 and/or B12.
* Planned cardiac, peripheral or cerebrovascular revascularization, defined as a decision taken by the patient and his or her physician(s) to perform surgical or percutaneous transluminal revascularization within the next 6 months.
* Hemodynamically significant primary valvular outflow tract obstruction (e.g. mitral stenosis, asymmetric septal hypertrophy, malfunctioning prosthetic valve).
* Constrictive pericarditis.
* Complex congenital heart disease.
* Syncopal episodes presumed to be due to uncontrolled life-threatening arrhythmias (asymptomatic arrhythmias including ventricular tachycardia are not exclusion criteria.
* Uncontrolled hypertension.
* Cor pulmonale.
* Heart transplant recipient.
* Other important non-cardiovascular disease(s) expected to limit compliance and/or impact on patient's ability to complete the study, such as: *history of alcohol or drug abuse, *psychiatric disorders, *senility, *severe physical disability, *illnesses including terminal stage of cancer and other major systemic illnesses expected to limit the patient's ability to comply with the study protocol and to complete the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000
Dates: Start 1999-12; Study Completion 2005-10

PRIMARY OUTCOMES:
The composite of cardiovascular death, myocardial infarction (MI) and stroke

SECONDARY OUTCOMES:
Total major ischemic events (includes CV [cardiovascular] death, MI, stroke, hospitalizations for UA [unstable angina] and revascularizations)
Hospitalization for unstable angina
Hospitalization for congestive heart failure (CHF)
Hospitalization for revascularization procedures
Total mortality
Other hospitalizations
Diabetic complications (laser therapy, dialysis, nephropathy or new diagnosis of diabetes)
The composite of death due to cancer, hospitalization for cancer and new diagnosis of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Lonn, MD MSc FRCPC FACC, Principal Investigator — McMaster University
Locations (1):
- McMaster University and Hamilton Health Sciences Corporation, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Saposnik G, Ray JG, Sheridan P, McQueen M, Lonn E; Heart Outcomes Prevention Evaluation 2 Investigators. Homocysteine-lowering therapy and stroke risk, severity, and disability: additional findings from the HOPE 2 trial. Stroke. 2009 Apr;40(4):1365-72. doi: 10.1161/STROKEAHA.108.529503. Epub 2009 Feb 19. PMID 19228852
- [Derived] Held C, Sumner G, Sheridan P, McQueen M, Smith S, Dagenais G, Yusuf S, Lonn E. Correlations between plasma homocysteine and folate concentrations and carotid atherosclerosis in high-risk individuals: baseline data from the Homocysteine and Atherosclerosis Reduction Trial (HART). Vasc Med. 2008 Nov;13(4):245-53. doi: 10.1177/1358863X08092102. PMID 18940900
- [Derived] Mann JF, Sheridan P, McQueen MJ, Held C, Arnold JM, Fodor G, Yusuf S, Lonn EM; HOPE-2 investigators. Homocysteine lowering with folic acid and B vitamins in people with chronic kidney disease--results of the renal Hope-2 study. Nephrol Dial Transplant. 2008 Feb;23(2):645-53. doi: 10.1093/ndt/gfm485. Epub 2007 Nov 14. PMID 18003666
- [Derived] Sawka AM, Ray JG, Yi Q, Josse RG, Lonn E. Randomized clinical trial of homocysteine level lowering therapy and fractures. Arch Intern Med. 2007 Oct 22;167(19):2136-9. doi: 10.1001/archinte.167.19.2136. No abstract available. PMID 17954810
- [Derived] Ray JG, Kearon C, Yi Q, Sheridan P, Lonn E; Heart Outcomes Prevention Evaluation 2 (HOPE-2) Investigators. Homocysteine-lowering therapy and risk for venous thromboembolism: a randomized trial. Ann Intern Med. 2007 Jun 5;146(11):761-7. doi: 10.7326/0003-4819-146-11-200706050-00157. Epub 2007 Apr 30. PMID 17470822
- [Derived] Lonn E, Yusuf S, Arnold MJ, Sheridan P, Pogue J, Micks M, McQueen MJ, Probstfield J, Fodor G, Held C, Genest J Jr; Heart Outcomes Prevention Evaluation (HOPE) 2 Investigators. Homocysteine lowering with folic acid and B vitamins in vascular disease. N Engl J Med. 2006 Apr 13;354(15):1567-77. doi: 10.1056/NEJMoa060900. Epub 2006 Mar 12. PMID 16531613
- See also: Population Health Research Institute - click on HOPE-TOO for more information about the study — http://www.phri.ca